CLINICAL TRIAL: NCT06330519
Title: "Impact of Different Techniques on the Efficacy of Anaesthesia in Mandibular Molars With Acute Irreversible Pulpitis: A Randomized Controlled Trial"
Brief Title: Enhancing Anaesthetic Success in Mandibular Molars With Symptomatic Irreversible Pulpitis: A Comparative Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ainshams University Dentistry
Record Dates: First submitted 2024-03-08; First posted 2024-03-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-03

CONDITIONS: Pulpitis - Irreversible
Keywords: dexamethasone; intraligamentary; cryotherapy
MeSH Terms: interventions — dexamethasone 21-phosphate; norflurane; Dental Pulp Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- intraligamentary dexamethazone (Experimental)
  Interventions: Drug: Dexamethasone sodium phosphate injection
- Endo-ice cryotherapy (Active Comparator)
  Interventions: Other: 1,1,1,2 tetrafluoroethane
- Intraoral soft tissue cryotherapy (Active Comparator)
  Interventions: Other: intraoral soft tissue cryotherapy
- Inferior Alveolar nerve block only (No Intervention)

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate injection — Patients receive 0.8ml of dexamethazone by periodontal ligament injection 30 minutes before the inferior alveolar nerve block
  Arms: intraligamentary dexamethazone
Other: 1,1,1,2 tetrafluoroethane — EndoIce (1,1,1,2 tetrafluoroethane) applied on the buccal, lingual (3 s/surface), and occlusal surfaces (4 s) for a total of 10 s then standard IANB was administered
  Other Names: Endo-ice
  Arms: Endo-ice cryotherapy
Other: intraoral soft tissue cryotherapy — Small ice packs (wrapped in sterile gauze) placed intraorally in the mouth on the vestibular surface of the treated tooth for 5 minutes then standard IANB was administered
  Arms: Intraoral soft tissue cryotherapy

SUMMARY:
The goal of this clinical trial is to assess the effect of

* Preoperative intraligamentary corticosteroids injection
* Cryotherapy which is cold application on :

  * Hard tooth structure ( crown of the tooth )
  * Soft tissue overlying roots on the efficacy of the inferior alveolar nerve block anaesthesia in patients with mandibular molars with symptomatic irreversible pulpitis. The main question it aims to answer are: • Does intraligamentary dexamethazone injection increase the success rate of inferior alveolar nerve block without the need for oral premedication.

Participants will describe their preoperative pain level to the investigator and describe their pain level during the treatment.

Researchers will compare cryotherapy to see if it increases the success rate of inferior alveolar nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to commit for the entire period of the trial and agreed to sign the written consent after full explanation of the study.
* Having a mandibular molar tooth diagnosed with symptomatic irreversible pulpitis (hot tooth - vital pulp, intermittent or continuous sharp pain that lasts longer after removal of the stimulus).

Exclusion Criteria:

* Presence of any systemic disease or allergic reactions.
* Vulnerable group; prisoners, pregnant females, mentally ill, etc…
* The presence of a periapical radiolucency.
* Teeth with open apices.
* A previous root canal treatment.
* Sinus tracts.
* Local gum swelling around the affected tooth.
* Severe periodontal disease .
* Presence of periodontal pockets >3 mm in the affected tooth.
* Absence of bleeding in the pulp chamber on access cavity preparation.
* Patients with doubted diagnosis due to multiple carious teeth.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
The effect of intraligamentary dexamethazone injection on the success rate of inferior alveolar nerve block | Assessed up to 30 minutes, from lip numbness point until the end of pulp extirpation.
  Percentage of the successful participants among total participants

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided